CLINICAL TRIAL: NCT02139540
Title: Nitrous Oxide as Treatment for Major Depression - a Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201204023
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Depression; Major Depressive Disorder
Keywords: Treatment
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Nitrous Oxide; Nitrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N2O/Placebo (Other): First session: Nitrous oxide Second session: placebo
  Interventions: Drug: Nitrous Oxide; Drug: Placebo
- Placebo/N2O (Other): First session: Placebo Second session: Nitrous Oxide
  Interventions: Drug: Nitrous Oxide; Drug: Placebo

INTERVENTIONS:
Drug: Nitrous Oxide — Patients will receive either up to 50% nitrous oxide/50% oxygen for 1 hour or "placebo" (50% nitrogen [inert]/50% oxygen) in two separate sessions. Both sessions will be 1 week apart.
  Other Names: Laughing Gas
Drug: Placebo — 50% nitrogen [inert]/50% oxygen - otherwise completely identical administration and setup
  Other Names: 50% nitrogen [inert]/50% oxygen

SUMMARY:
Major depressive disorder (MDD) is a global medical problem with significant shortcomings in current therapy. Chief among these is the delay between initiation of pharmacologic therapy and clinical improvement in symptoms. Recently ketamine, an NDMA-receptor antagonist has been shown to rapidly and effectively reverse the symptoms of MDD. Nitrous oxide, another NMDA-receptor antagonist, may produce the same effect with a cleaner side-effect profile and perhaps without the need for intravenous access and anesthesia personnel. Therefore, we propose conducting a pilot randomized placebo controlled double-blind crossover study in which patients will receive up to 50% nitrous oxide in oxygen or up to 50% oxygen in air for a period of one hour in addition to standard medical therapy. Depression severity will be assessed by a blinded observer pre-treatment, 30 minutes and 2 hours post treatment using the Hamilton depression rating scale.

DETAILED DESCRIPTION:
We will study 20 patients with non-treatment resistant major depression and 20 patients with treatment-resistant major depression, defined as failure of at least 2 antidepressants in the current depressive episode and 3 lifetime medication failures.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18-65 years of age
2. Major depressive disorder without psychosis with as determined by structured interview using the Mini-International Neuropsychiatric Interview (MINI).

   (baseline )
3. HDRS-21 score of >18
4. Good command of the English language

Exclusion Criteria:

History of:

1. Bipolar disorder
2. Schizoprenia
3. Schizoaffective disorder
4. Obsessive-compulsive disorder, panic disorder
5. Substance abuse or dependence (except for remote substance abuse or dependence with remission at least 1 year prior to the study and except for nicotine use disorders)
6. Axis II diagnoses that may interfere with the patient's ability to improve on nitrous oxide
7. Acute medical illness that may pose subject at risk during nitrous oxide administration
8. Active suicidal intention (inability to contract for safety)
9. Active psychotic symptoms
10. Patients with significant pulmonary disease and/or requiring supplemental oxygen
11. Contraindication against the use of nitrous oxide:

    1. Pneumothorax
    2. Bowel obstruction
    3. Middle ear occlusion
    4. Elevated intracranial pressure
    5. Chronic cobalamin and/or folate deficiency treated with folic acid or vitamin B12
    6. Pregnant patients
    7. Breastfeeding women
12. Previous administration of NMDA-receptor antagonists (e.g., ketamine) within the last 3 months
13. Current electro-convulsive therapy treatment
14. Any active suicidal ideation, intention, or planning (clinical assessment of suicidality will be used)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nagele, MD, MSc, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] de Leon VC, Kumar A, Nagele P, Palanca BJ, Gott B, Janski A, Zorumski CF, Conway CR. Nitrous Oxide Reduced Suicidal Ideation in Treatment-Resistant Major Depression in Exploratory Analysis. J Clin Psychiatry. 2023 Aug 16;84(5):22br14725. doi: 10.4088/JCP.22br14725. No abstract available. PMID 37585253

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 Participants were consented, however only 20 continued.
Period: Overall Study
Arm/Group | N2O/Placebo | Placebo/N2O
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N2O/Placebo | Placebo/N2O | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [30 to 55] | 48 [30 to 55] | 48 [30 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Rating Scale HDRS-21
Description: (21-point Hamilton Depression Rating Scale) Scoring is based on the first 17 items on the 21 point scale. Eight items are scored on a 5-point scale, ranging form 0=not present to 4= severe. Nine are scored from 0-2.
Time Frame: baseline and 24 hours
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Nitrous Oxide | Placebo
Number analyzed (Participants) | 20 | 20
score on a scale | 5.5 [2.5 to 8.5] | 2.8 [0.2 to 5.8]
Statistical Analysis 1: Comparison: Nitrous Oxide vs Placebo; The primary outcome (HDRS-21) was analyzed with a repeated-measures mixed effects linear model using restricted maximum likelihood estimation. To adjust for the observed carryover effect, the model included a randomization group term and a three-way interaction (treatment × time × randomization group); Test type: Superiority; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Change in Quick Inventory of Depressive Symptomatology - Self Report - QIDS -SR
Description: [Quick Inventory of Depressive Symptomatology - Self Report] An item-by-item severity scale of 0 to 3, with possible total scores ranging from 0 to 84. The items on the scale are added together for a total score. Higher scores mean worse outcome.
Time Frame: baseline and 24 hours
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Nitrous Oxide | Placebo
Number analyzed (Participants) | 20 | 20
score on a scale | 3.2 [1.3 to 5.0] | 1.0 [0.9 to 2.8]
Statistical Analysis 1: Comparison: Nitrous Oxide vs Placebo; Test type: Superiority; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 2 Weeks
Arm/Group | Nitrous Oxide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 14/20 | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nitrous Oxide (N=20) | Placebo (N=20)
Nausea and Vomiting (Gastrointestinal disorders) | 3 | 0
Headache (Nervous system disorders) | 2 | 2
Dizziness (General disorders) | 1 | 2
Numbness (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Panic Attack (Psychiatric disorders) | 1 | 0
Claustrophobia (Psychiatric disorders) | 1 | 0
Hyperventilation (General disorders) | 1 | 0
Regurgitation (Gastrointestinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes